CLINICAL TRIAL: NCT05130073
Title: The Role of a 4-point Therapy Response Score With PET/CT Post Definitive Chemoradiation for Anal Squamous Cell Cancer: A Prospective Study
Brief Title: 4-Point Therapy Response Score With PET/CT for Anal Squamous Cell Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA19-0088; NCI-2021-10964 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA19-0088 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-12

CONDITIONS: Anal Squamous Cell Carcinoma; Stage 0 Anal Cancer AJCC v8; Stage I Anal Cancer AJCC v8; Stage II Anal Cancer AJCC v8; Stage IIA Anal Cancer AJCC v8; Stage IIB Anal Cancer AJCC v8; Stage III Anal Cancer AJCC v8; Stage IIIA Anal Cancer AJCC v8; Stage IIIB Anal Cancer AJCC v8; Stage IIIC Anal Cancer AJCC v8
MeSH Terms: conditions — Anus Neoplasms | interventions — Chromatin Immunoprecipitation Sequencing; Follow-Up Studies; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (PET/CT, medical data review, follow-up): Patients undergo PET/CT at baseline and at 3 months post therapy completion. Patients' medical records are received. Patients are followed up for 5 years.
  Interventions: Procedure: Computed Tomography; Other: Electronic Health Record Review; Procedure: Follow-Up; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Electronic Health Record Review — Review of medical records
Procedure: Follow-Up — Undergo follow-up
  Other Names: Active Follow-up; Clinical Signs Follow-up; CLSFUP; Follow Up; follow_up; Followed; Followup
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This study determines whether a positron emission tomography (PET)/computed tomography (CT) 4-point scoring system may predict overall survival for anal squamous cell cancer patients. A 4-point scoring system involving imaging scans may help to predict how patients with anal squamous cell cancer respond to chemoradiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether a PET/CT scoring system in invasive biopsy proven anal squamous cell carcinoma (SCCA) to be treated with chemoradiation with curative intent (any T any N) predicts for overall survival (OS).

SECONDARY OBJECTIVES:

I. To determine whether a PET/CT scoring system in invasive biopsy proven SCCA to be treated with definitive chemoradiation with curative intent predicts for progression free survival (PFS).

II. To determine and validate inter-reader reliability. III. To calculate C-index to evaluate the prognostic capacity of PET/CT scores for survival.

IV. To determine the association between pre-treatment PET/CT scores after treatment and OS.

EXPLORATORY OBJECTIVE:

I. To correlate level of standardized uptake value (SUV) pre and post therapy and its correlation with overall survival.

OUTLINE:

Patients undergo PET/CT at baseline and at 3 months post therapy completion. Patients' medical records are received. Patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed biopsy proven invasive SCCA (any T, any N) deemed a candidate to undergo standard of care definitive chemoradiation at MD Anderson Cancer Center (MDACC) with curative intent
* Age > 18 years at time of study entry
* Ability to provide written informed consent

Exclusion Criteria:

* Patients unwilling to participate in a PET/CT at baseline and at 3 months post completion of definitive chemoradiation
* Patients with an active second primary malignancy requiring chemotherapy or radiation treatment
* Stage IV SCCA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with invasive SCCA
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Through study completion, an average of 1 year
  The Kaplan-Meier method will be used. Log rank test will be used to compare OS between positron emission tomography (PET)/computed tomography (CT) negative and positive tumor group. Multivariable Cox proportional hazards models will be fitted to evaluate the association between OS and PET/CT scores, adjusting for the effects of covariates. In addition to positive and negative tumor groups, PET/CT scores of 4 categories will also be analyzed. C-index will be calculated to evaluate the prognostic capacity of PET/CT score with survival outcomes. Additionally, the Cohen kappa coefficient will be calculated to measure inter-reader agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Benny Johnson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org